CLINICAL TRIAL: NCT01471860
Title: Neo Randomized Heart Failure Study
Brief Title: BAROSTIM NEO System in the Treatment of Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360029
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device and Medical Management (Experimental): Medical Management, to be determined by the participant's physician, described as:
  * Optimal pharmacological therapy: Prescribed to a beta blocker, a diuretic, and an ACE (Angiotensin-converting-enzyme) inhibitor or ARB (Angiotensin Receptor Blocker) unless contraindicated or not tolerated. These drugs must be used in a manner consistent with their labeling.
  * Stable pharmacological therapy: No more than a 50% increase or a 50% decrease of the dosage of any one medication, and post titration of all heart failure medications.
  Participants should remain on their prescribed heart failure medications and same dosing schedule for the duration of the study unless investigators determine medically necessary changes are needed. Additionally, every effort should be made to maintain adequate rate control for subjects with atrial fibrillation throughout the duration of the study.
  Interventions: Device: BAROSTIM NEO System; Drug: Medical Management

INTERVENTIONS:
Device: BAROSTIM NEO System
  Other Names: XR-1 System; Neo System
Drug: Medical Management

SUMMARY:
The purpose of this portion of study NCT01471860 is to assess the long-term safety and efficacy of the BAROSTIM NEO System in Canadian study participants implanted with the device.

DETAILED DESCRIPTION:
The Neo Randomized Heart Failure Study is a prospective, randomized, study describing the safety and efficacy of the BAROSTIM NEO System in the heart failure participants with a left ventricular ejection fraction ≤ 35%.

During long-term follow-up, all participants are required to have at least one annual visit.

Parameters assessed during long-term follow-up visits:

* Physical Assessment
* Subject Medications
* Serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Actively participating in the Neo Randomized Heart Failure Study.
* Have signed a revised approved informed consent form for continued participation in this study.

Exclusion Criteria:

* Treating physician decision that the subject should not continue with therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2021-08-11 (Estimated)

PRIMARY OUTCOMES:
To assess long-term adverse events in Canadian participants implanted with the BAROSTIM NEO System | For the duration of the study, up to 5 years.
  Ascertain the type, frequency, severity and timing of long-term adverse events in participants implanted with the device, while providing a viable treatment option to participants currently implanted with the BAROSTIM NEO System.

CONTACTS AND LOCATIONS:
Overall Officials: Uta Hoppe, MD, Principal Investigator — University of Cologne
Locations (30):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta - Edmonton, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Montreal Heart Institute, Montreal, Quebec
- France (3):
  - CHRU de Lille, Lille
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse
- Germany (17):
  - Vivantes Hospital Berlin, Berlin
  - Immanuel Hospital Bernau-Heart Center Brandenburg, Bernau
  - University Hospital Cologne, Cologne
  - University Hospital Essen, Essen
  - CVC Frankfurt, Frankfurt
  - University Hospital Giessen, Giessen
  - Georg August University - Goettingen, Göttingen
  - Klinik St. Georg, Hamburg, Hamburg
  - University Heart Center Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital of Schleswig-Holstein, Kiel Campus, Kiel
  - Klinikum St. Georg Leipzig, Leipzig
  - Klinikum Ludenscheid, Lüdenscheid
  - University Hospital Mannheim, Mannheim
  - Lukas Hospital Neuss, Neuss
  - Oldenburg Hospital, Oldenburg
  - Reinbek Hospital, St. Adolf-Stift, Reinbek
- Italy (5):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Opedali, Ancona
  - Azienda Ospedaliera Spedali Riuniti Di Bergamo, Bergamo
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Istituto Scientifico San Luca, Milan

REFERENCES:
- [Result] Abraham WT, Zile MR, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):487-496. doi: 10.1016/j.jchf.2015.02.006. Epub 2015 May 14. PMID 25982108
- [Derived] Halbach M, Abraham WT, Butter C, Ducharme A, Klug D, Little WC, Reuter H, Schafer JE, Senni M, Swarup V, Wachter R, Weaver FA, Wilks SJ, Zile MR, Muller-Ehmsen J. Baroreflex activation therapy for the treatment of heart failure with reduced ejection fraction in patients with and without coronary artery disease. Int J Cardiol. 2018 Sep 1;266:187-192. doi: 10.1016/j.ijcard.2018.04.075. Epub 2018 Apr 21. PMID 29705650
- [Derived] Zile MR, Abraham WT, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex activation therapy for the treatment of heart failure with a reduced ejection fraction: safety and efficacy in patients with and without cardiac resynchronization therapy. Eur J Heart Fail. 2015 Oct;17(10):1066-74. doi: 10.1002/ejhf.299. Epub 2015 Jun 10. PMID 26011593